CLINICAL TRIAL: NCT00002344
Title: Double-Blind Crossover Study Assessing the Dose Proportionality of Azithromycin Tablets in HIV-Infected Subjects
Brief Title: A Study of Azithromycin in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 226C; 066-060
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Bacterial Infections; HIV Infections
Keywords: Azithromycin; Bacterial Infections
MeSH Terms: conditions — Bacterial Infections; HIV Infections | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
To assess the dose proportionality of azithromycin concentrations and toleration when delivered in tablet formulation to HIV-infected patients.

The need exists to further assess the antibacterial agent azithromycin at differing doses in an HIV-infected population.

DETAILED DESCRIPTION:
The need exists to further assess the antibacterial agent azithromycin at differing doses in an HIV-infected population.

Patients are randomized to receive azithromycin at 1 of 2 doses in a two-treatment, two-period, cross-over study. Dosing visits are separated by at least 14-day wash-out periods.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV seropositivity.
* CD4 count <= 500 cells/mm3.
* NO active AIDS opportunistic infection.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Other active intercurrent illness.
* Any condition possibly affecting drug absorption (e.g., ulcers, gastrectomy, HIV-associated enteropathies.
* Signs or symptoms of severe illness that would preclude study participation.
* Known allergies to macrolide antibiotics.

Patients with the following prior condition are excluded:

Clinically important change in baseline status within 4 weeks prior to study entry.

Prior Medication:

Excluded:

* Investigational drugs including treatment IND drugs within 4 weeks prior to study entry.

Known drug or alcohol dependence.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12

CONTACTS AND LOCATIONS:
Locations (1):
- Harris Laboratories Inc, Phoenix, Arizona, United States